CLINICAL TRIAL: NCT07269028
Title: Personalised and Gamification-based Decision Aid (DA): a Randomized Controlled Pilot Study About Colorectal Cancer (CRC) Screening
Acronym: DA-CRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Collaborators: Agenzia di Tutela della Salute (ATS) di Brescia (Unknown)
Responsible Party: Principal Investigator, Cristina Montomoli, Full Professor, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Protocol Number: NP5686
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Colo-rectal Cancer
Keywords: Colo-rectal cancer; Prevention; eHealth; Gamification
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Gamified Mobile App
- Control (No Intervention)

INTERVENTIONS:
Other: Gamified Mobile App — The intervention app included questionnaires on family history, knowledge of primary and secondary prevention, and locus of control (LoC), as well as gamification and reward features.
  Arms: Intervention

SUMMARY:
Colorectal cancer (CRC) is the second leading cause of cancer-related mortality worldwide, accounting for approximately 903,000 deaths annually. While population-based screening programmes have demonstrated effectiveness in enhancing early detection and reducing mortality, participation rates remain suboptimal. Adherence is influenced by cognitive, psychological, and socioeconomic barriers.

This study aimed to assess the impact of a digital decision aid (DA), incorporating personalisation and gamification elements, on informed decision-making and adherence to CRC screening.

DA-CRC is a two-arm randomised controlled pilot trial. Individuals born in 1973-1974 living in the area served by the local health authority of Brescia (Northern Italy) who were invited for the first time to participate in the CRC screening programme, were eligible. An invitation letter, including instructions to download the PREVenGO app, was mailed to potential participants.

Upon download, participants were randomised to either the intervention or control arm. The intervention app included questionnaires on family history, knowledge of primary and secondary prevention, and locus of control (LoC), as well as gamification and reward features. The control app provided static educational content only. Notifications prompted users to complete follow-up assessments at 3 months (T1) and 6 months (T2), receive prevention information, and attend screening.

ELIGIBILITY:
Inclusion Criteria:

* Stable residence within one of the municipalities served by Brescia LHA;
* Ownership of a smartphone (Android or iOS);
* Proficiency in the Italian language;
* Provision of informed consent within the PREVenGO app.

Exclusion Criteria:

* Failure to provide informed consent.

Ages: 50 Years to 51 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 248 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Awareness | From enrollment to 6 months
  Informed choice, using the three-dimensional model by Marteau, including:
  Knowledge (minimum score 7/13); Attitude (score >24); Behavioural intention (actual participation).

SECONDARY OUTCOMES:
Uptake of CRC screening | From enrollment to 31st December 2024
  ATS Brescia provided pseudonymised data on actual FOBT participation.
Knowledge of primary prevention and healthy behaviours, | From enrollment to 6 months
  Assessment through 13 multiple-choice questions. Participants were classified based on correct responses as:
  Low knowledge (0-5 correct answers); Moderate knowledge (6-8); High knowledge (9-13);
Decisional conflict, user satisfaction, and app acceptability | From enrollment to 6 months
  Evaluation through items related to the decision-making process and perceived usefulness of the decision aid

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Montomoli, Principal Investigator — University of Pavia
Locations (1):
- Agenzia per la Tutela della Salute (ATS) di Brescia, Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hersch J, Barratt A, Jansen J, Irwig L, McGeechan K, Jacklyn G, Thornton H, Dhillon H, Houssami N, McCaffery K. Use of a decision aid including information on overdetection to support informed choice about breast cancer screening: a randomised controlled trial. Lancet. 2015 Apr 25;385(9978):1642-52. doi: 10.1016/S0140-6736(15)60123-4. Epub 2015 Feb 18. PMID 25701273
- [Background] Wallston KA, Wallston BS, DeVellis R. Development of the Multidimensional Health Locus of Control (MHLC) Scales. Health Educ Monogr. 1978 Spring;6(2):160-70. doi: 10.1177/109019817800600107. PMID 689890
- [Background] Duan Y, Shang B, Liang W, Du G, Yang M, Rhodes RE. Effects of eHealth-Based Multiple Health Behavior Change Interventions on Physical Activity, Healthy Diet, and Weight in People With Noncommunicable Diseases: Systematic Review and Meta-analysis. J Med Internet Res. 2021 Feb 22;23(2):e23786. doi: 10.2196/23786. PMID 33616534
- [Background] Sequi-Dominguez I, Alvarez-Bueno C, Martinez-Vizcaino V, Fernandez-Rodriguez R, Del Saz Lara A, Cavero-Redondo I. Effectiveness of Mobile Health Interventions Promoting Physical Activity and Lifestyle Interventions to Reduce Cardiovascular Risk Among Individuals With Metabolic Syndrome: Systematic Review and Meta-Analysis. J Med Internet Res. 2020 Aug 31;22(8):e17790. doi: 10.2196/17790. PMID 32865503
- [Background] Mohamad Marzuki MF, Yaacob NA, Bin Yaacob NM, Abu Hassan MR, Ahmad SB. Usable Mobile App for Community Education on Colorectal Cancer: Development Process and Usability Study. JMIR Hum Factors. 2019 Apr 16;6(2):e12103. doi: 10.2196/12103. PMID 30990454
- [Background] Hammedi, W., Leclerq, T. & Van Riel, A. C. R. The use of gamification mechanics to increase employee and user engagement in participative healthcare services: A study of two cases. J. Serv. Manag. 28, 640-661 (2017).
- [Background] Rotter, J. B. (1954). Social learning and clinical psychology. Prentice-Hall, Inc
- [Background] Roberto A, Colombo C, Candiani G, Satolli R, Giordano L, Jaramillo L, Castagno R, Mantellini P, Falini P, Carnesciali E, Valenza M, Costa L, Campari C, Caroli S, Faggiano RC, Orione L, Belmessieri B, Marchio V, Deandrea S, Silvestri A, Luciano D, Paci E, Mosconi P. A dynamic web-based decision aid to improve informed choice in organised breast cancer screening. A pragmatic randomised trial in Italy. Br J Cancer. 2020 Sep;123(5):714-721. doi: 10.1038/s41416-020-0935-2. Epub 2020 Jun 17. PMID 32546834
- [Background] Gabel P, Larsen MB, Edwards A, Kirkegaard P, Andersen B. Effectiveness of a decision aid for colorectal cancer screening on components of informed choice according to educational attainment: A randomised controlled trial. PLoS One. 2020 Nov 10;15(11):e0241703. doi: 10.1371/journal.pone.0241703. eCollection 2020. PMID 33170877
- [Background] Stacey D, Legare F, Lewis K, Barry MJ, Bennett CL, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Thomson R, Trevena L. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2017 Apr 12;4(4):CD001431. doi: 10.1002/14651858.CD001431.pub5. PMID 28402085
- [Background] Elwyn G, Frosch D, Rollnick S. Dual equipoise shared decision making: definitions for decision and behaviour support interventions. Implement Sci. 2009 Nov 18;4:75. doi: 10.1186/1748-5908-4-75. PMID 19922647
- [Background] O'Connor AM, Legare F, Stacey D. Risk communication in practice: the contribution of decision aids. BMJ. 2003 Sep 27;327(7417):736-40. doi: 10.1136/bmj.327.7417.736. PMID 14512487
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-03-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT07269028/Prot_SAP_ICF_000.pdf